CLINICAL TRIAL: NCT00784394
Title: Phase I Ascending Single Dose Pharmacokinetics (PK) and Safety Study of 3,3' Di-indolylmethane (DIM)
Brief Title: Diindolylmethane in Preventing Cancer in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2014-00523; NCI-2014-00523 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NO1-CN-35008-38; CDR0000617334; KUMC-HSC-9139 (Other: University of Kansas Medical Center); N01-CN-35008-1 (Other: DCP); N01CN35008 (NIH)
Record Dates: First submitted 2008-11-01; First posted 2008-11-04 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — 3,3'-diindolylmethane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (diindolylmethane) (Experimental): Participants receive a single dose of diindolylmethane PO on day 1.
  Interventions: Drug: diindolylmethane; Other: pharmacological study; Other: laboratory biomarker analysis; Other: quality-of-life assessment
- Arm II (placebo) (Placebo Comparator): Participants receive a single dose of placebo orally (PO) on day 1.
  Interventions: Other: placebo; Other: pharmacological study; Other: laboratory biomarker analysis; Other: quality-of-life assessment

INTERVENTIONS:
Drug: diindolylmethane — Given PO
  Other Names: DIM
  Arms: Arm I (diindolylmethane)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase I clinical trial studies the side effects and best dose of diindolylmethane in preventing cancer in healthy volunteers. Diindolylmethane is formed in the stomachs of people who eat a chemical that is normally found in vegetables, including cabbage, broccoli, Brussels sprouts, cauliflower, and watercress. Diindolylmethane may prevent the development of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine single oral doses of 3,3' di-indolylmethane (DIM) (diindolylmethane) that are safe and well- tolerated.

II. To determine the pharmacokinetics of these single oral doses of DIM.

OUTLINE: This is a dose-escalation study. Participants are randomized to 1 of 2 treatment arms.

ARM I: Participants receive a single dose of diindolylmethane orally (PO) on day 1.

ARM II: Participants receive a single dose of placebo orally (PO) on day 1.

After completion of study treatment, participants are followed up on days 2, 3, and 6.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers and non-users of abuse drugs as confirmed by urine cotinine (Accutest NicoMeter Urine Professional strip or equivalent test) and drug screen at visit 1
* Free of acute, unstable, chronic or recurring medical conditions based on history, physical examination, laboratory tests; the laboratory tests to be performed will be: blood serum chemistry screen to include comprehensive metabolic panel (glucose, creatinine, urea nitrogen [blood urea nitrogen (BUN)], sodium, potassium, chloride, calcium, total bilirubin, protein, albumin, globulin, cholesterol and the enzymes alkaline phosphatase, aspartate aminotransferase [AST], and alanine aminotransferase [ALT]) and lipid panel (total, low density lipoprotein [LDL] and high density lipoprotein [HDL] cholesterol and triglycerides); complete blood count including differential and platelet count; prothrombin time; and routine urinalysis; values for laboratory tests must be within the ranges below grade 2 of Common Toxicity Criteria (CTC) and/or as specified below:
* Hemoglobin > 10 g/dL
* Absolute granulocyte count > 1500/ìL
* Creatinine < 2.0 mg/dl
* Albumin > 3.0 g/dl
* Bilirubin < 1.8 mg/dl
* AST < 110 U/l
* ALT < 110 U/l
* Alkaline phosphatase < 300 U/l
* Subjects must weigh +/- 20% of ideal body weight by the Metropolitan Life tables
* Men or women who are strict vegetarians or who eat more than 3 medium servings (1/2 cup each) of cruciferous vegetables per week will be excluded; those who stop ingesting cruciferous vegetables >= 14 days and alcohol >= 7 days before starting DIM and agree to refrain from taking them for the duration of the study will not be excluded; cruciferous vegetables include broccoli, cabbage (including coleslaw), cauliflower, bok-choy, Brussels sprouts, collards, kale, kohlrabi, mustard greens, rutabaga, turnip, and watercress; participants will be asked to complete a brief diet questionnaire listing these vegetables to assess these criteria; caffeine- and grapefruit-containing foods and beverages are to be avoided for at least 48 hours before visit 2 (DIM dosing)

Exclusion Criteria:

* Subjects with serious drug allergies or other serious intolerance or allergies will be excluded; those with mild seasonal allergies will be accepted
* Subjects with chronic headaches, dysphoria, fatigue, dizziness, blurred vision, insomnia, rhinorrhea, nausea, vomiting, abdominal pain, diarrhea, constipation, or similar conditions
* Subjects with a serious acute or chronic illness (diabetes, arthritis, asthma, etc.) or requiring chronic drug therapy, who continuously take supplements or have taken an investigational drug within the past three months
* Subjects who have evidence of an active malignancy or have received chemotherapy, and/or antiestrogen therapy
* Subjects who have a life expectancy of < 12 months
* Subjects who have regularly taken over the past 21 days any concomitant medications, herbal products, dietary supplements or vitamins; women taking oral contraceptives will be accepted; women who are pregnant (positive urine human chorionic gonadotropin [hCG] at visit 2) or lactating will be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD), defined as the highest dose at which no grade 2 or higher toxicities are seen | Up to day 6
  Frequencies and percents will be used to summarize the toxicities seen at each dose level and overall. Descriptive statistics will be calculated on all variables of interest: frequencies and percentages will be used to summarize categorical variables and medians, and ranges will summarize quantitative variables.

SECONDARY OUTCOMES:
Pharmacokinetics of diindolylmethane | Baseline and at 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours after administration
  Pharmacokinetic parameters such as half-life, maximum concentration (Cmax), time of Cmax (Tmax), and area under the concentration-time curve (AUC) will be calculated for all subjects who complete the study. It is anticipated that a one-compartment elimination model will fit the data. These parameters will be summarized at each dose and overall with median and ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Aryeh Hurwitz, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States